CLINICAL TRIAL: NCT05990049
Title: Impact of Hyaluronic Acid on Free Gingival Graft Healing and Palatal Donor Site Wound Healing
Brief Title: Hyaluronic Acid and Free Gingival Graft Healing
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Zagreb (Other)
Responsible Party: Principal Investigator, Ana Badovinac, assistant professor, University of Zagreb
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 05-PA-30-V-2/2022.
Record Dates: First submitted 2023-07-03; First posted 2023-08-14 (Actual); Last update posted 2023-08-16 (Actual); Status verified 2023-08

CONDITIONS: Hyaluronic Acid; Gingival Recession, Localized; Pain, Postoperative
Keywords: keratinized tissue width; shrinkage; hyaluronic acid; free gingival graft
MeSH Terms: conditions — Gingival Recession; Pain, Postoperative

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Hyaluronic acid (Active Comparator): During the surgery, the hyaluronic acid will be administered on donor site wound and on recipient site before suturing.
  Interventions: Drug: Hyadent BG
- Control (No Intervention): After the harvesting of the graft from the donor site, the wound will be sutured using only saline to clean the wound.
  On the recipient site, before positioning the graft, only saline will be used.

INTERVENTIONS:
Drug: Hyadent BG — Hyadent BG is a cross-linked hyaluronic acid. 1,6% cross-linked hyaluronic acid (xHA), 0,2% native hyaluronic acid (HA)
  Arms: Hyaluronic acid

SUMMARY:
This study aims to evaluate the impact of locally applied hyaluronic acid on free gingival graft wound bed healing and palatal donor site wound healing.

Forty subjects will be randomly divided in two separate groups. Test group will be treated with hyaluronic acid during the procedure and the control group without.

Periodontal parameters and other clinical measurements will be taken on baseline, 7 days postoperative, 14 days postoperative, 1 month, 3 months and 6 months postoperative.

DETAILED DESCRIPTION:
Free gingival graft is common, simple and predictable surgical procedure. Patients who have keratinized tissue width less than 2 mm will undergo the surgery after passing the inclusion criteria together with initial periodontal therapy. Total number of 40 patients will be divided in two separate groups; test group (hyaluronic acid) and control group based on random choice.The randomization will be examiner blind.

After the application of local anaesthesia, surgical procedure will be done in the same groups equally. In the recipient site, an horizontal incision will be performed on the mucogingival junction or 1-2 mm above it to include the free marginal gingiva. Partial thickness flap will be dissected in order to ensure the vascularisation of the graft. The size of the incision and graft will depend on the keratinized tissue width of the teeth area.

The graft will be taken from the donor site on the anterior palate in the area of premolars and molars. The graft will be measured with periodontal probe (UNC-15) in 3 dimensions over the flat surface and after the harvesting will be put in glass with saline. Donor site will be sutured using fibrin sponge and non-resorbable sutures. The size of recipient site and graft will depend on number of teeth with keratinized tissue width less than 2 mm.

The graft will be positioned on the recipient site and stabilised using non-resorbable suture performing single sutures and a sling suture around the tooth. The group of patients who will receive the hyaluronic acid will be treated on donor and recipient site before the suturing, applied once on the wound bed.

Postoperatively, patients will be instructed to rinse with 0.12% chlorhexidine digluconate twice a day. The patients will be asked to keep a diary for 7 days about pain sensations using VAS scale for donor and recipient site. An analgetic treatment will be prescribed if needed.

Recall visits will be 7 and 14 days postoperatively. The 7th day postoperatively will be removed sutures from donor site, and on 14th day the sutures from the graft and recipient site.

Clinical measurements with periodontal indices will be taken on 1, 3, and 6 months follow up.

ELIGIBILITY:
Inclusion Criteria:

* no systemic disease
* healthy
* non-smokers
* at least one tooth with keratinized tissue width less than 2 mm

Exclusion Criteria:

* heavy smokers
* younger than 18years old
* using drugs
* allergy on anesthesia
* using drugs or alcohol
* undergoing chemotherapy
* undergoing radiotherapy

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2023-03-01 (Actual); Primary Completion 2024-01-01 (Estimated); Study Completion 2024-03-01 (Estimated)

PRIMARY OUTCOMES:
Keratinized tissue gain | baseline to 1 month postoperatively
  changes of the tissue in apico - coronal dimensions from gingival margin to mucogingival junction
Keratinized tissue gain | baseline to 3 months postoperatively
  changes of the tissue in apico - coronal dimensions from gingival margin to mucogingival junction
Keratinized tissue gain | baseline to 6 months postoperatively
  changes of the tissue in apico - coronal dimensions from gingival margin to mucogingival junction
Shrinkage of the graft | baseline to 1 month postoperatively
  changes of the graft in apico - coronal and mesio-distal dimensions
Shrinkage of the graft | baseline to 3 months postoperatively
  changes of the graft in apico - coronal and mesio-distal dimensions
Shrinkage of the graft | baseline to 6 months postoperatively
  changes of the graft in apico - coronal and mesio-distal dimensions

SECONDARY OUTCOMES:
Dimensional changes in gingival recessions | baseline to 1 month postoperative
  reduction of gingival recessions
Dimensional changes in gingival recessions | baseline to 3 months postoperative
  reduction of gingival recessions
Dimensional changes in gingival recessions | baseline to 6 months postoperative
  reduction of gingival recessions

CONTACTS AND LOCATIONS:
Overall Officials: Ana Badovinac, assoc prof, Study Director — School of Dental Medicine University of Zagreb
Locations (1):
- School of Dental Medicine University of Zagreb, Zagreb, Croatia

IPD SHARING:
Plan to Share IPD: No